CLINICAL TRIAL: NCT02635737
Title: Safety and Feasibility Study of Magnetic Seed Markers to Localise Breast Cancers for Surgical Excision
Brief Title: Magnetic Seed Localisation of Breast Cancers
Acronym: Sentimark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Endomagnetics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016BR005
Record Dates: First submitted 2015-11-16; First posted 2015-12-21 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sentimark device placement (Experimental): Sentimark device placed in women having mastectomy surgery
  Interventions: Device: Sentimark

INTERVENTIONS:
Device: Sentimark — Placement of a metallic clip with paramagnetic properties for tumour localisation

SUMMARY:
This is a single site, single arm, unblinded safety and feasibility cohort study investigating the use of magnetic marker seeds to localise breast tumours.

DETAILED DESCRIPTION:
Background and Rationale Breast Cancer Breast cancer is a heterogeneous disease, with great diversity in the site, size and progression of tumours. Some are palpable and discovered by the patient, though many are first detected during mammogram screening. For such cancers, localisation is necessary prior to surgery, to guide surgeons to the target excision site.

Wire Guided Localisation Traditionally, localisation involves radiographic-guided insertion of a wire into the breast, with positioning of the wire tip at the centre of the lesion. However, this procedure carries several logistical limitations , stemming from the fact that wire localisation must be performed on the day of surgery. This is to minimise risk of wire migration or dislodgement , a significant possibility due to the external section of wire left protruding from the breast. Same-day appointments demand excellent coordination between radiological departments and operating theatres to ensure that disruption to procedure scheduling is minimised. Delays may result from technically difficult procedures , leading to over-running radiology appointments that have a knock on effect on operating lists. Additionally, cancelled operations can result in preceding wire guidance procedures becoming unnecessary, resulting in wasted staff hours.

Another limitation of wire guidance occurs because the wire directs surgeons along a linear route. Lesions are found at a point along the wire, though it can be difficult to determine how far along they are found. For this reason, surgeons making initial incisions may be dictated by the visual trajectory of the wire, rather than the location of the lesion. This can lead to excessive dissection and sub optimal cosmetic results.

Radioactive Seed Localisation Radioactive seed localisation (RSL) is a localisation technique that is less commonly used in the United Kingdom (UK). A radioactive seed can be inserted up to 5 days before surgery, thus eliminating the requirement for radiology appointments on the same day as the patient's operation. The seed is detected in theatre using a handheld gamma probe. The gamma probe directs the surgeon to a single specific point via the shortest route, whereas, wires often transect the breast, meaning that surgeons commonly end up dissecting across normal tissue to locate the tip of the wire. In addition, with RSL, there is no distraction from external projections of wire, so the surgeon is guided purely by the audible response to the seed. It is hypothesised that the advantages of RSL will lead to improved surgical techniques and reduce pressures on theatre scheduling.

However, up to now, there is little evidence demonstrating clear superiority in surgical outcome of one localisation technique. Several studies have found lower positive margin rates in patients undergoing RSL versus wire guidance , , . This means that edges of excised tissues less commonly involves cancerous tissue, suggesting that RSL more accurately localises cancerous lesions. Conversely, many more studies, including one of the largest trials to date, conclude there is no variability in surgical outcome.

Regardless of stance on surgical outcome, all studies noted that RSL offers significant improvements in scheduling of appointments and patient convenience.

However, radioactive techniques are not without limitations. Several studies have evaluated the use of standard radioisotope and blue dye injections for sentinel node biopsy. Each study commented on the complex legislation regulating use of radioisotopes, particularly with regards to operator training and correct disposal and handling. In addition, radioisotope use increases patient and healthcare worker radiation exposure which, though minimal, would be preferable to avoid.

Iron Oxide Use in Breast Surgery Several studies have investigated the use of liquid injections of iron oxide rather than traditional radioisotope and blue dye injections, in sentinel node identification. Following iron oxide injections, a handheld magnetometer was used to detect the location of iron oxide in the lymph nodes. All studies concluded that iron oxide particles performed equally as well as standard radioisotope & blue dye injections in sentinel node identification, demonstrating potential for more widespread use of the technique.

In addition, Ahmed et al tested localisation of cancerous lesions using a magnetic tracer injection. The tracer successfully localised all tumours and resulted in appropriate excisional margins, without excess tissue excision; thus demonstrating the feasibility of magnetic tracer localisation of tumours.

Sentimark Magnetic Localisation The localisation method with which this project is concerned has similar principles to RSL. However, instead of radioactive seeds, a soft magnetic seed called Sentimark, is placed into the breast. The seed is similar to a biopsy clip and can be detected using a handheld magnetometer called Sentimag. The Sentimag probe emits an alternating magnetic field that detects the magnetic response of the Sentimark seed. The magnetometer produces an audible response when held close to the Sentimark seed and can be used by surgeons to locate target excision sites. Sentimark is inserted about a week before operation, ideally during a biopsy appointment, for patient convenience.

This study will be the first to investigate magnetic seed localisation of tumours. It is hypothesised that using magnetic seeds rather than injections with a magnetic tracer will allow more accurate detection and localisation using the Sentimag probe. This is because the probe is detecting the magnetic field produced by a single discrete object, rather than a collection of iron oxide-containing liquid which may disperse throughout the breast.

Summary of Localisation Techniques The coordination and scheduling difficulties encountered in wire guided localisation, alongside the logistical and safety issues of radioisotope usage, highlight a requirement for further innovation and acquisition of new technologies in the field of localisation. It is hoped that magnetic seed localisation can act as a feasible alternative to existing technologies. Use of magnetism in localisation techniques offers a potential alternative to wire guidance and RSL.

An important consideration with the deployment of the new seed is whether the size and shape of the seed are sufficiently similar to previous designs to show similar migration patterns, as movement of the seed prior to surgery can cause incomplete lesion excision with en-suing requirements for re-operation or an increased risk of recurrence.

The migration performance of Sentimark in an implantation trial in goats, mean migration of 1.1mm with a range 0 to 3.6mm (N=10), was very similar to that observed by Alderliesten, et al. who report a mean migration of 0.8mm, range 0 to 2.8mm (N=10) for RSL seeds which was considered "clinically negligible" in RSL of human breast lesions. However, confirmation is required that the magnetic marker performs as expected in the clinic.

The study will test a soft magnetic seed (Sentimark) and its accompanying handheld magnetic probe (Sentimag) with particular consideration for its safety and performance once placed into human breast tissue.

Device The device to be studied is a small (5mm x 0.9mm) metal magnetic marker (seed) that has soft magnetic properties. This means that when exposed to a magnetic field it becomes magnetic. The magnetism can then be detected using a magnetometer and probe which gives an audible and visual signal of the strength of response from the seed and as it is directional this can accurately guide the user to the site of the magnetic seed. The magnetometer is a CE (Conformite Europeene) approved device and is used worldwide for detecting iron oxide in sentinel lymph node biopsy procedures, and is proven in clinical practice. The seed itself will be deployed by a radiologist into the centre of the tumour site using a similar technique to that used to currently place a wire into the breast. The seed itself is cylindrical and in in vivo studies in goats have shown similar migration performance to that seen with radioactive seeds in human breast tissue.

The seed has also been tested in animal tissue models by (University Hospital of South Manchester) UHSM radiologists and surgeons, and in these models it can be safely deployed by the radiologists using existing techniques. The device was detected and surgical resection was performed with 100% accuracy on all specimens. There is no radiation exposure from this device.

Study Population Adult women with capacity to consent who have a proven breast cancer requiring breast removing mastectomy surgery.

Potential Risks to Patients The device itself is a small piece of metal and in itself does not offer a likely safety risk.

* Migration of the seed - the seed is cylindrical and therefore once placed in the breast it has the potential to migrate along the path of the needle that was used to deploy it. When deployed into mammary soft tissue in animal models the device has not migrated. This study will involve placing the device in women having mastectomy so even if the device migrates it will not affect patients cancer care (as the whole breast will be removed along with the device no matter where it is located in the breast);
* Failure to detect the seed - the seed is small and the magnetic field generated is proportional to the size of the seed. This study aims to assess whether the seed can be detected in all sizes of breast as in some cases it may be possible that the seed lies too deep in the breast to be detected using the magnetometer. To ensure safe resection of the cancer, each patient in this study will be under-going a planned mastectomy, to ensure that the device is fully removed even if detection should fail;
* Tissue acceptance - the seed is produced from a single material and has demonstrated biocompatibility through ISO-10993 biocompatibility evaluation including demonstration of tissue acceptance in mammary tissue of goats (28-day implantation period). Bone wax is used as a terminal plug for Sentimark device. Bone wax is commonly used for the same purpose in brachytherapy and RSL needles. Some reaction to bone wax may occur, such as an allergic reaction or foreign body reactions (e.g. granulomas), as bone wax is a minimally resorbable implantable substance.

Potential Benefits The study will be carried out in patients requiring a mastectomy. In this population, the full cycle of marker (seed) deployment and removal can be evaluated, but as the breast is being removed as part of the planned cancer treatment, patient treatment will be unaffected should the magnetic seed not perform as intended. However, there will be no direct benefit for patients taking part in the study and the potential benefits of this study are limited to the advancement of medical knowledge. If the study confirms that the magnetic marker (seed) is safe and the method is feasible, the device has the potential to be used for localisation of breast cancers for lumpectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study;
* Female, aged 18 years or above;
* Diagnosed with breast cancer (invasive or dcis);
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study;
* Undergoing mastectomy breast surgery.

Exclusion Criteria:

* Patients with a Pacemaker or implanted device;
* Patients requiring an MRI scan prior to surgery;
* Patients with known coagulopathy or receiving anticoagulant medication including warfarin, heparin, clopidogrel or rivaroxaban;
* Patients receiving Neoadjuvant chemotherapy;
* Patients who are pregnant or lactating;
* Patients scheduled for immediate breast reconstruction;
* Patients who have received Sienna (iron oxide) injection in the previous six months;
* Patients with an existing breast haematoma close to the target lesion.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Harvey, MBBS PhD, Principal Investigator — University Hospital of South Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sentimark Device Placement
Started | 29
Completed | 28
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Females having mastectomy surgery
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 54 [37 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 28
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Migration of Sentimark Device
Description: Migration of the device>10mm between mammograms, clip position >40mm from target lesion
Time Frame: 1-4 weeks from placement
Population: migration of seed
Measure: Number; unit: percentage of Magseed migrating >10mm
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
percentage of Magseed migrating >10mm | 100

2. Secondary Outcome: Accuracy of Initial Placement
Description: distance of the marker (seed) on radiographic imaging from the intended site of placement (e.g. lesion, marker clip, calcification) in mm
Time Frame: within 60 minutes of seed placement
Measure: Mean (Standard Error); unit: mm
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
mm | 0 (0.1)

3. Secondary Outcome: Percentage Magnetic Markers (Seeds) Within Target Area;
Description: The target area will be detected by mammography on the day of surgery and is defined as within 10mm of the target lesion
Time Frame: within 60 minutes of seed placement
Population: all 28 womens markers were within the target area
Measure: Number; unit: percentage of womens markers were within
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
percentage of womens markers were within | 100

4. Secondary Outcome: Depth of Marker (Seed)
Description: Marker (seed) depth to the nearest skin surface will be estimated sonographically in mm
Time Frame: within 60 minutes of seed placement
Measure: Mean (Full Range); unit: mm
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
mm | 16 [3.5 to 30]

5. Secondary Outcome: Number of Seeds Detectable on the Sentimag Detector
Description: ability to detect the marker (seed) with Sentimag - this will be recorded whether the count is detectable on the Sentimag detector
Time Frame: Within 60 minutes of seed placement
Measure: Count of Participants; unit: Participants
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
Participants | 28

6. Secondary Outcome: Host Response to Implanted Seed Device
Description: percentage of seeds showing foreign body reaction histopathologically
Time Frame: within 4 weeks of seed placement
Measure: Number; unit: percentage of seeds showing fb reaction
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 18
percentage of seeds showing fb reaction | 50

7. Other Pre Specified Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: The number of treatment related adverse and serious adverse events will be recorded as a number of events and a percentage of participants who experienced an Adverse Event
Time Frame: Through study completion, an average of six weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
Participants | 0

8. Other Pre Specified Outcome: Mastectomy Weight
Description: Mastectomy weight - breast weight
Time Frame: At Surgery
Population: breast weight
Measure: Mean (Full Range); unit: grams
Arm/Group | Sentimark Device Placement
Number analyzed (Participants) | 28
grams | 833 [126 to 2600]

ADVERSE EVENTS:
Time Frame: six weeks perioperatively
Description: standard descriptions
Arm/Group | Sentimark Device Placement
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT02635737/Prot_SAP_000.pdf